CLINICAL TRIAL: NCT05658510
Title: Efficacy And Safety of BXCL501 Evaluated For At-Home Use In A Multisite Double-Blind Placebo-Controlled Trial For Agitation Associated With Schizophrenia And Bipolar Disorder
Brief Title: Dexmedetomidine in the Treatment of Agitation Associated With Schizophrenia and Bipolar Disorder (SERENITY III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXCL501-401
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Agitation,Psychomotor; Bipolar I Disorder; Bipolar II Disorder; Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Psychomotor Agitation; Bipolar Disorder; Schizophrenia; Psychotic Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Part 1: Patients randomized to receive 60 mcg of BXCL501 or a matching placebo.
  Part 2: Patients randomized to receive 120 mcg of BXCL501 or a matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: 60 mcg of BXCL501 (Experimental): Sublingual film containing 60 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Part 1: Matching Placebo (Placebo Comparator): Sublingual Placebo film
  Interventions: Drug: Matching Placebo
- Part 2: 120 mcg of BXCL501 (Experimental): Sublingual film containing 120 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Part 2: Matching Placebo (Placebo Comparator): Sublingual Placebo film
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BXCL501 — Sublingual Film
  Other Names: Dexmedetomidine
  Arms: Part 1: 60 mcg of BXCL501; Part 2: 120 mcg of BXCL501
Drug: Matching Placebo — Sublingual Placebo Film
  Other Names: Placebo
  Arms: Part 1: Matching Placebo; Part 2: Matching Placebo

SUMMARY:
In this study, an investigational medication named BXCL501 is being tested for the treatment of episodes of agitation associated with bipolar I and bipolar II disorder, schizophrenia, schizoaffective and schizophreniform disorder. This study compares the study drug to a placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2-Part, Phase III study to assess the efficacy, safety, and tolerability of BXCL501 in adult (18-75 years old) males and females with agitation episodes associated with a primary diagnosis of bipolar I disorder, bipolar II disorder, schizophrenia, schizoaffective disorder, or schizophreniform disorder. Part 1 of the study is a one-day, in-clinic treatment of 60 mcg dose, and post-treatment observation period with patients experiencing an acute episode of agitation. Part 1 is now complete. Part 2 of the study is a 12-week study to determine the safety of a BXCL501 120 mcg dose when used as needed for episodes of agitation at home.

ELIGIBILITY:
A patient may enroll in only one part of the study; either Part 1 or Part 2.

Inclusion Criteria:

* Male and female patients between the ages of 18 to 75 years, inclusive
* Patients who can read, understand and provide written informed consent.
* Patients who have met Diagnostic and Statistical Manual5/5-Text Revision criteria for bipolar I or bipolar II disorder, schizophrenia, schizoaffective or schizophreniform disorder.
* Patients who, in the opinion of the Principal Investigator, are in good general health before study participation based on a detailed medical history, a physical examination, a 12-lead ECG, a blood chemistry profile, hematology, and urinalysis.
* Participants who agree to use a medically acceptable and effective birth control method

Part 1 only

* Patients who are judged to be clinically agitated at Screening and Baseline with a total score of ≥ 14 on the 5 items (poor impulse control, tension, hostility, uncooperativeness, and excitement) comprising the PEC.
* Patients with a score of ≥4 on at least 1 of the 5 items on the PEC at Baseline.

Part 2 only

* Patients have had at least three clinical presentations of agitation requiring an intervention (e.g., receipt of as needed [PRN] medication for the episode, clinic visit, emergency room visit, emergency medical services intervention, law enforcement intervention) in the past three months prior to Screening
* Patients who are receiving stable psychotropic treatment for 30 days prior to Screening for the underlying primary diagnosis and who are expected to remain on stable treatment for the duration of the study.
* The patient can understand and follow the study procedures, including completing the Agitation Episode Diary.

Exclusion Criteria:

* Patients with serious or unstable medical illnesses. These include current hepatic (moderate-severe hepatic impairment), renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease, congestive heart failure), endocrinologic, or hematologic disease.
* A history of agitation episodes due to substance use.
* A diagnosis of antisocial personality disorder, borderline personality disorder, or narcissistic personality disorder that predated the diagnosis of schizophrenia or bipolar disorder
* Patients who are judged to be at significant risk of suicide
* Female patients who have a positive pregnancy test at Screening or Baseline, or are breastfeeding.
* Patients currently treated with alpha-1 noradrenergic blockers (terazosin, doxazosin, tamsulosin, alfuzosin, or prazosin), alpha-2 adrenergic agonists, or other prohibited medications.
* Patients with hydrocephalus, seizure disorder, or history of significant head trauma, stroke, transient ischemic attack, subarachnoid bleeding, brain tumor, encephalopathy, meningitis, Parkinson's disease, or focal neurological findings.
* History of syncope or other syncopal attacks, current evidence of hypovolemia, or orthostatic hypotension
* Patients with laboratory or ECG abnormalities considered clinically significant by the Investigator
* Patients who have received an investigational drug within 30 days before the study start
* Patients who have previously received BXCL501 via prescription (under the trade name IGALMI™) or received BXCL501 in clinical trial
* Patients considered by the Investigator to be unsuitable candidates for receiving dexmedetomidine or considered to be unsuitable for participating in the study for any reason.

Part 1 only

* Patients with agitation caused by acute intoxication, including identification of alcohol by breathalyzer or drugs of abuse (except for THC) during urine screening.
* Use of benzodiazepines or other hypnotics or antipsychotic drugs in the 4 hours before study treatment.

Part 2 only

* Psychiatric comorbidities are generally allowed; however, moderate or severe substance use disorders (SUD) (within the past 6 months) are exclusionary if the substance involved is other than nicotine or caffeine. Cannabis use is not exclusionary if it is not the focus of treatment in the last 6 months before Screening.
* Self-injurious behavior that is active.
* Patients with known personal or family history of genetic long QT syndrome.

Informant Inclusion Criteria:

* At least 18 years of age at the time of screening.
* Is a spouse, significant other, family member, friend, or home health aide, residence manager of an adult patient who is determined to be eligible for the study per the patient inclusion/exclusion criteria.
* Has known the patient for at least 3 months cumulatively.
* Currently living with or routinely contacting the patient at least five days a week.
* Does not plan to discontinue contact with the patient during the study period.
* Willing and able to provide written informed consent.
* Willing and able to follow the study procedures, including completing the Agitation Episode Diary and other study procedures during the study.
* Willing and able to accompany patient and remain present at the clinical site during the clinic visits and be interviewed by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Change from baseline in Positive and Negative Syndrome Scale - Excited (PEC) total score | 2 hours
  The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)
Part 2: The incidence of SAEs and TEAEs compared with placebo. | Through study completion, an average of 12 weeks
  To assess the safety of 120 mcg BXCL501 when used in an at-home environment based on serious adverse events (SAE) and treatment emergent adverse events (TEAEs).

SECONDARY OUTCOMES:
Part 1: Clinical Global Impression - Improvement (CGI-I) | 2 hours
  The Clinical Global Impression - Improvement (CGI-I) for agitation in response to treatment measures the current level of agitation relative to the level of agitation prior to administration of study intervention. The CGI-I scores range from 1 to 7 with a score of 1 indicating very much improved, and a score of 7 indicating very much worse.
Part 1: Change in Modified Clinical Global Impression - Severity (mCGI-S) scores from Baseline | 2 hours
  The Modified Clinical Global Impression - Severity (mCGI-S) measures the current level of agitation. For this study, the mCGI-S is a 4-point scale where a score of 0 represents no agitation, and scores of 1-3 describe increasing severities of agitation (mild, moderate, severe).
Part 1:The number of responders based on the Modified Clinical Global Impression - Severity (mCGI-S) score | 2 hours
  The Modified Clinical Global Impression - Severity (mCGI-S) measures the current level of agitation. A responder is characterized as a participant with a score of 0 (represents no agitation) or 1 (mild agitation)
Part 1:Change from baseline in Agitation-Calmness Evaluation Scale (ACES) | 2 hours
  The Agitation-Calmness Evaluation Scale (ACES) is a single item scale that measures overall agitation and sedation, where a score of 1 indicates marked agitation; 2 - moderate agitation; 3 - mild agitation; 4 - normal behavior; 5 - mild calmness; 6 - moderate calmness; 7 - marked calmness; 8 - deep sleep; and 9 - unarousable.
Part 1: Incidence of treatment-emergent adverse events (TEAEs) | Through study completion, an average of 8 hours
  To assess the safety of BXCL501 based on treatment-emergent adverse events (TEAEs)
Part 1: Change from baseline in heart rate (HR) at rest | Baseline, and 2, 4, 6, and 8 hours postdose
  The effect of BXCL501 on heart rate at rest
Part 1: Change from baseline in heart rate (HR) under orthostatic stress | Baseline, and 2, 4, 6, and 8 hours postdose
  The effect of BXCL501 on heart rate under orthostatic stress
Part 1: Change from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) at rest | Baseline, and 2, 4, 6, and 8 hours postdose
  The effect of BXCL501 on systolic and diastolic blood pressure at rest
Part 1: Change from baseline in systolic blood pressure (SBP) and diastolic blood pressure (DBP) under orthostatic stress | Baseline, and 2, 4, 6, and 8 hours postdose
  The effect of BXCL501 on systolic and diastolic blood pressure under orthostatic stress
Part 1: Incidence of abnormal electrocardiograms (ECG) reported as an adverse event (AE) | Through study completion, an average of 8 hours
  Any abnormal ECG value that is reported as an adverse event (AE)
Part 1: Incidence of abnormal clinical laboratory values reported as an adverse event (AE) | Through study completion, an average of 8 hours
  Any abnormal clinical laboratory value that is reported as an adverse event (AE)
Part 2: Incidence of interactions with emergency services related to agitation | Through study completion, an average of 12 weeks
  Evaluate the impact of BXCL501 on the use of healthcare and emergency service resources because of agitation episodes
Part 2: Incidence of overall adverse events and AEs leading to discontinuation | Through study completion, an average of 12 weeks
  To evaluate the safety and tolerability profile of 120 mcg BXCL501

CONTACTS AND LOCATIONS:
Overall Officials: Matt Mandel, MD, Study Chair — BioXcel Therapeutics
Locations (24):
- United States (24):
  - BioXcel Clinical Research Site 113, Bellflower, California
  - BioXcel Clinical Research Site 128, Cerritos, California
  - BioXcel Clinical Research Site 110, Culver City, California
  - BioXcel Clinical Research Site 108, Garden Grove, California
  - BioXcel Clinical Research Site 117, Lemon Grove, California
  - BioXcel Clinical Research Site 121, Los Angeles, California
  - BioXcel Clinical Research Site 123, Oceanside, California
  - BioXcel Clinical Research Site 104, Orange, California
  - BioXcel Clinical Research Site 133, Rancho Cucamonga, California
  - BioXcel Clinical Research Site 114, Riverside, California
  - BioXcel Clinical Research Site 129, Denver, Colorado
  - BioXcel Clinical Research Site 131, Miami, Florida
  - BioXcel Clinical Research Site 124, Miami, Florida
  - BioXcel Clinical Research Site 130, Elgin, Illinois
  - BioXcel Clinical Research Site 103, Gaithersburg, Maryland
  - BioXcel Clinical Research Site 118, Las Vegas, Nevada
  - BioXcel Clinical Research Site 137, Las Vegas, Nevada
  - BioXcel Clinical Research Site 105, Berlin, New Jersey
  - BioXcel Clinical Research Site 122, Beachwood, Ohio
  - BioXcel Clinical Research Site 136, Austin, Texas
  - BioXcel Clinical Research Site 102, DeSoto, Texas
  - BioXcel Clinical Research Site 125, Irving, Texas
  - BioXcel Clinical Research Site 127, Plano, Texas
  - BioXcel Clinical Research Site 126, Everett, Washington

IPD SHARING:
Plan to Share IPD: No